CLINICAL TRIAL: NCT05609526
Title: Target Muscles Training in Patients With Leg Lymphedema : Inspiratory Muscles Versus Calf Muscles
Brief Title: Inspiratory and Calf Muscles Training in Patients With Leg Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ilknur Mazı, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC-AKGUL-001
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Lymphedema of Leg; Lymphedema; Exercise
Keywords: Diagragma; Calf Muscle
MeSH Terms: conditions — Lymphedema; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1.Group (Compression Therapy) (No Intervention): The patient will be placed in the supine position. Short stretch bandages of 6, 8, 10 and 12 cm will be applied to the extremity in a multi-layered and special way. Starting with the finger bandage, the pressure will be reduced as it goes distally. The patient's gait and circulation will be checked after bandaging is finished.
  will be.
- 2.Group (Inspiratory muscle training) (Experimental): Maximum inspiratory intraoral pressure (MIP) and expiratory intraoral pressure (MEP) will be measured before patients begin IMT. Total training time 30 minutes per day will be. On the first day, the MIP levels of the participants will be evaluated and the training workload will be determined as 30% of the MIP. For IMT, after a nose clip was inserted from the participants They will be asked to sit on the mouthpiece of the device and close their lips tightly. With the device in this position, the device for four to five breath rests after every 10 breathing cycles.
  mouth, and repeat the cycle for 15 minutes.
  Interventions: Other: Compression Therapy; Other: Inspiratory muscle training
- 3.Group (Calf muscle exercise training) (Experimental): A strengthening treatment program will be applied to the calf muscles. CMET will consist of static stretching exercise for the dorsiflexors and plantar flexors, isotonic resistance exercise with elastic resistance bands, heel and toe lift in both feet, followed by toe raising and lowering without heel raising. An isotonic exercise (mini squat) will be performed for ankle pumping exercise and knee flexion in sitting position. Patients will begin strength training with elastic resistance bands using red bands (lowest resistance). Green and blue bands by increasing the number of sets and repetitions will start to be used (increased resistance). (31.32)
  Interventions: Other: Compression Therapy; Other: Calf muscle exercise training
- 4.Group (Inspiratory and calf muscle training) (Experimental): All applications made in 3 groups will be made in this group.
  Interventions: Other: Compression Therapy; Other: Inspiratory muscle training; Other: Calf muscle exercise training

INTERVENTIONS:
Other: Compression Therapy — 6, 8, 10 and 12 cm short tension bandages multi-layered and will be applied specifically to the extremity. Starting with the finger bandage, the pressure will be reduced as it goes distally.
  Arms: 2.Group (Inspiratory muscle training); 3.Group (Calf muscle exercise training); 4.Group (Inspiratory and calf muscle training)
Other: Inspiratory muscle training — Maximum inspiratory intraoral pressure (MIP) and expiratory intraoral pressure (MEP) will be measured before patients begin IMT. Total training time per day will be 30 minutes.
  Arms: 2.Group (Inspiratory muscle training); 4.Group (Inspiratory and calf muscle training)
Other: Calf muscle exercise training — A strengthening treatment program will be applied to the calf muscles.dorsiflexors and plantar flexors will consist of static stretching exercise, isotonic resistance exercise with elastic resistance bands, heel and toe raising in both feet, followed by toe raising and lowering without raising the heel.
  Arms: 3.Group (Calf muscle exercise training); 4.Group (Inspiratory and calf muscle training)

SUMMARY:
Lymphedema results in the accumulation of protein-rich fluid in the subcutaneous tissue as a result of the failure of the lymphatic system, which returns water and protein in the interstitial spaces to the bloodstream. The aim of its treatment is to return this fluid accumulated in the interstitial space to the venous system. Early diagnosis and subsequent treatment of lymphedema, which is a chronic and progressive problem, is important to improve symptoms and prevent complications. Exercises recommended by specialist physiotherapists increase lymph flow and improve protein resorption. Exercises applied with compression bandages or compression garments provide significant improvement in patients with lymphedema.

The aim of this study is to provide inspiratory muscle training and leg compression therapy together with compression therapy in patients with lower extremity lymphedema.

To evaluate the effectiveness of these exercises on the patient's extremity volume and fullness, tissue water content, edema status, walking capacity, functionality and quality of life by comparing the effectiveness of muscle exercise training. In addition, researchers aim to determine the more effective exercise method for these patients.

DETAILED DESCRIPTION:
Lymphedema is a chronic, progressive disease that occurs with the accumulation of protein-rich fluid in the interstitial tissue spaces as a result of abnormal development or damage to the lymphatic system. Exercise is one of the components of Complex Relief Physiotherapy, which is used as the gold standard in the treatment of lymphedema. exercises put pressure on lymphatic vessels with rhythmic contraction and relaxation of muscle groups. Thus, smooth muscle contraction in the lymphatic vessels is triggered. The transport of lymph fluid is possible with the activation of the muscles that provide the movement of the skin. It has been shown that strengthening the calf muscle with exercise can improve the pumping function, increase the average peak torque of the muscle, decrease the severity of the disease, increase the ankle joint movement, increase the calf muscle endurance and improve the quality of life. The pump power of the inspiratory muscles is also important in the lymph circulation, as well as in the venous circulation.

This study will include 45 patients who volunteered to participate in the study, who were treated at Istanbul University- Cerrahpasa Faculty of Health Sciences and Gerontology Research and Application Center from October 2022 to October 2023. Lymphedema Quality of Life Scale for Evaluation (LYQOL) Lower Extremity Perimeter Measurement Numerical Rating Scale . 6 Minute Walk Test. Tissue Dielectric Constant (TDC) will be used.

Participants will be randomly divided into 4 groups. Only compression therapy(CT) will be given to the 1st group, inspiratory muscle training (IMT) in addition to the compression therapy to the 2nd group, and Calf muscle exercise training to the 3rd group in addition to CT.

CT will be applied to the patients in all four groups for 45-60 minutes a day, 6 days a week, for 4 weeks. Patients in the other 2 groups will participate in an exercise program for 4 weeks, 4 days a week, in addition to CT. The power analysis will be calculated based on the 5% margin of error, 95% confidence level, using the Raosoft sample size and the clinically significant minimum difference of LYMQOL, one of the primary measurement tools.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with lymphedema
* No visual or hearing impairment
* Being literate in Turkish
* 18- 75 years old

Exclusion Criteria:

* Acute infection
* Aardiac edema
* Peripheral arterial diseases
* Congestive advanced heart failure
* Malignant lymphedema
* Having a psychiatric disorder requiring prior vessel ablation and/or prescription medication
* Having a neurological, orthopedic or rheumatological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-11-14 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-09-12 (Estimated)

PRIMARY OUTCOMES:
Lymphedema Quality of Life Scale | 5 minute
  Evaluates the effect of arm and leg edema on quality of life with separate questionnaires.
  It consists of 4 subscales: function, appearance, symptom and mood. The score of each item ranges from 1 to 4 (1 = not at all, 2 = a little, 3 = a lot, 4 = a lot). The score of each scale is calculated by dividing the total score by the number of items and ranges from 1 to 4. It is concluded that the higher the score, the more the quality of life is affected.
Lower Extremity Perimeter Measurement | 5 minute
  It will be calculated using the Frustum Formula from circumference measurements taken at 10 cm intervals from the tip of the second toe to the thigh. Patients' affected and unaffected lower extremities will be measured with standard fiberglass. Measurements will be made by the same physiotherapist before and after the 4-week intervention.

SECONDARY OUTCOMES:
Numerical Rating Scale | 5 minute
  Subjective feedback of patients regarding leg fullness associated with lymphedema will be recorded by the scoring method of the affected lower extremity. This scoring will be between 0 and 10.
6-Minute Walk Test | 10minute
  It is used to determine walking capacity by measuring the maximum distance an individual can walk in six minutes.
Tissue Dielectric Constant (TDC) | 5 minute
  The tissue dielectric constant (TDC) technique gives information about the emergence of lymphedema in the early stages and the change in the amount of water under the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Akgül, Study Director — dean at university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sander AP, Hajer NM, Hemenway K, Miller AC. Upper-extremity volume measurements in women with lymphedema: a comparison of measurements obtained via water displacement with geometrically determined volume. Phys Ther. 2002 Dec;82(12):1201-12. PMID 12444879
- [Background] Kocak Z, Overgaard J. Risk factors of arm lymphedema in breast cancer patients. Acta Oncol. 2000;39(3):389-92. doi: 10.1080/028418600750013168. PMID 10987236
- [Background] Gashev AA. Physiologic aspects of lymphatic contractile function: current perspectives. Ann N Y Acad Sci. 2002 Dec;979:178-87; discussion 188-96. doi: 10.1111/j.1749-6632.2002.tb04878.x. PMID 12543727
- [Background] Olszewski WL. Contractility patterns of human leg lymphatics in various stages of obstructive lymphedema. Ann N Y Acad Sci. 2008;1131:110-8. doi: 10.1196/annals.1413.010. PMID 18519964
- [Background] Browse NL. The pathogenesis of venous ulceration: a hypothesis. J Vasc Surg. 1988 Mar;7(3):468-72. doi: 10.1067/mva.1988.avs0070468. No abstract available. PMID 3346962
- [Background] Szuba A, Rockson SG. Lymphedema: anatomy, physiology and pathogenesis. Vasc Med. 1997 Nov;2(4):321-6. doi: 10.1177/1358863X9700200408. PMID 9575606
- [Background] Aydin G, Yeldan I, Akgul A, Ipek G. Effects of inspiratory muscle training versus calf muscle training on quality of life, pain, venous function and activity in patients with chronic venous insufficiency. J Vasc Surg Venous Lymphat Disord. 2022 Sep;10(5):1137-1146. doi: 10.1016/j.jvsv.2022.04.012. Epub 2022 Jun 14. PMID 35710091
- [Background] Do JH, Kim W, Cho YK, Lee J, Song EJ, Chun YM, Jeon JY. EFFECTS OF RESISTANCE EXERCISES AND COMPLEX DECONGESTIVE THERAPY ON ARM FUNCTION AND MUSCULAR STRENGTH IN BREAST CANCER RELATED LYMPHEDEMA. Lymphology. 2015 Dec;48(4):184-96. PMID 27164764
- [Background] Keeley V. Quality of life assessment tools in chronic oedema. Br J Community Nurs. 2008 Oct;13(10):S22-7. doi: 10.12968/bjcn.2008.13.Sup5.31193. PMID 19057479
- [Background] Solari E, Marcozzi C, Negrini D, Moriondo A. Lymphatic Vessels and Their Surroundings: How Local Physical Factors Affect Lymph Flow. Biology (Basel). 2020 Dec 11;9(12):463. doi: 10.3390/biology9120463. PMID 33322476
- [Derived] Akgul A, Mazi I, Aydin G, Yavuz M, Yeldan I. The effect of muscles in the treatment of lower limb lymphedema: respiratory muscles or leg muscles? Support Care Cancer. 2025 Apr 11;33(5):375. doi: 10.1007/s00520-025-09436-3. PMID 40214771